CLINICAL TRIAL: NCT04695561
Title: Investigation of the Effects of Different Myofascial Release Techniques on Pain, Functionality and Performance in Athletes With Iliotibial Band Tightness
Brief Title: Effects of Different Myofascial Release Techniques on Iliotibial Band Tightness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KaratayUSonmezTez
Record Dates: First submitted 2020-11-19; First posted 2021-01-05 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2020-11

CONDITIONS: Fascia Lata
Keywords: Fascia Lata; Fascia; Massage; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self Myofascial Relaxation (Experimental): In addition to the exercises applied to the participants in the control group, the participants in this group used Foam Roller, which was performed with the principle of painless movement 2 times a week for a total of 12 times a week for 6 weeks.
  Interventions: Other: Self Myofascial Relaxation
- Instrument Assisted Soft Tissue Mobilization (Experimental): In addition to the exercises applied to the participants in the control group, the participants in this group used Instrument Assisted Soft Tissue Mobilization, which was performed with the principle of painless movement 2 times a week for a total of 12 times a week for 6 weeks.
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization
- Only Exercise (Control) (Active Comparator): Stretching and strengthening exercises for the hip flexors, hip extensors and iliotibial band were shown to the participants in the control group for 6 weeks every day of the week.
  Interventions: Other: Only Exercise (Control)

INTERVENTIONS:
Other: Self Myofascial Relaxation — Total of 12 times for 6 weeks
  Arms: Self Myofascial Relaxation
Other: Instrument Assisted Soft Tissue Mobilization — Total of 12 times for 6 weeks
  Arms: Instrument Assisted Soft Tissue Mobilization
Other: Only Exercise (Control) — Every day for 6 weeks
  Arms: Only Exercise (Control)

SUMMARY:
The aim of the study is to investigate the effects of foam roller and instrument assisted soft tissue mobilization on pain, functionality and performance in athletes with iliotibial band tightness

DETAILED DESCRIPTION:
Subject In this study, the effects of foam roller myofascial massage and instrument assisted soft tissue mobilization (IASTM) (massage performed by applying light pressure to the skin with a tool) on pain, functionality and performance will be investigated in athletes with iliotibial band tightness. There are studies on both IASTM and Foam Roller Massage in the literature and they are popular applications recently. However, within our knowledge, when we look at the Turkish and English literature, no study has been found that compares these two therapeutic massages in terms of pain, functionality and performance.

Purpose Poor posture, facial traumas and stiffness cause tension in the fascia of that region and result in pain. This disrupts the complementary mechanism of the fascia, causing the structures attached to the fascia to be out of the normal sequence. Facial problems have an important place in athletes. Facial problems cause pain in the athlete, reducing the athlete's sportive performance and negatively affecting their functionality. In order to prevent these limitations and accelerate the recovery, the rehabilitation process is started after the surgery. Various exercises and myofascial massages are routinely applied to problems seen in athletes. Myofascial massage techniques can be used in athletes' problems for many positive reasons such as effective in a short time, rapid results, high success rate, risk-free and painless if experts do. Thanks to the findings to be obtained from our study, it is aimed to contribute to the literature with objective, evidence-based results in this field.

ELIGIBILITY:
Inclusion Criteria:

* The leg inclinations of the athletes evaluated with the Ober test will be measured with an inclinometer and the athletes below 25 degrees will be included in the study.
* Age between 18 and 30 years
* Agree to participate in the study,

Exclusion Criteria:

• Not having surgery

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-03-14 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Isokinetic Strength at 6 weeks | [Baseline and 6 weeks]
  It is a very effective force work since the muscles are dynamically loaded at their maximum capacity at all points of the angle of motion during isokinetic contraction. In our study, hip flexor-extensor, hip abductor-adductor, knee flexor-extensor muscle strength will be evaluated with the humac norm 2004 cybex isokinetic device.
Change from baseline in Pain Threshold Score at 6 weeks | [Baseline and 6 weeks]
  Pressure pain threshold is expressed as the lowest pressure giving pain or discomfort. "J Tech Commander Algometer" will be used to evaluate the pain threshold in our study. The device is a digital pain threshold measuring device and 1 cm. It consists of a sensor connected to a diameter hard tip. Pain in individuals with iliotibial band tension is 3 cm above the femur lateral condyle. The participant will be asked to stop the measurement by warning the therapist as soon as the pressure turns into a painful feeling. the minimum values mean worse outcome the maximum values mean better outcome
Change from baseline in Vertical Jump Distance at 6 weeks | [Baseline and 6 weeks]
  Vertical jump test will be used to measure the lower extremity explosive power of the subjects. A digital Jump Meter will be used to measure the vertical jump distance of the subjects. Before the test, the subjects will be allowed enough trials to reach the maximal height. For the test, subjects will be asked to stand on the Jump Meter's mat. Subjects will be instructed to jump to the greatest possible distance with both feet, allowing their arms and feet to swing. After the splash, they should land on the mat as a double foot. The test will be repeated 3 times, a 1-minute rest interval will be given between tests and the best grade will be recorded in cm
Change from baseline in Pro-Agility Test at 6 weeks | [Baseline and 6 weeks]
  The test called pro-agility will be used. At the starting point, the athlete will spread his legs, turn with the command to start and run fast to the right, touching the line 5 yards (4.6m) away with his right hand. The athlete will then turn left, quickly running to the ground 10 yards (9.1 m) away and touching the far line with his left hand. The athlete will turn back from the right and quickly run 5 yards between the start and the finish line, and the test will be completed.
Change from baseline in Postural Control at 6 weeks | [Baseline and 6 weeks]
  Postural control performances of the athletes will be determined by the Balance Error Scoring System. The original name of the test is Balance Error Scoring System (BESS) and it has been translated into Turkish as Balance Error Scoring System. Test, subjects 20 sec. They are required to maintain their test positions under 6 different conditions, eyes closed and without any support: flat and foam surface and 3 separate stance positions (double leg, single leg and tandem). A gym floor will be used for the flat surface. For the foam surface, a medium density foam block of 50x41x6 cm will be used (Airex Balance Pad, Alcan Airex AG, CH-5643 Sins / Switzerland)
Change from baseline in Modified Star Balance Test at 6 weeks | [Baseline and 6 weeks]
  Modified Star Balance Test is a method adapted from the Star Excursion Balance Test, which originally evaluated reaching in eight different directions, and is used in balance assessment. Extension directions were reduced to three as anterior, posteromedial and postero-lateral. The inter-rater and intra-rater reliability of Modified Star Balance Test was found to be quite high (95% CI: 0.88-0.99 p <0.01)
Change from baseline in Range of Motion (ROM) Assessment at 6 weeks | [Baseline and 6 weeks]
  ROM of the lower extremities will be evaluated with a goniometer.
Change from baseline in Lower extremity functional scale (LEFS) at 6 weeks | [Baseline and 6 weeks]
  It is a patient-reported questionnaire that evaluates the functional status of patients with musculoskeletal dysfunction affecting their lower extremities. The questionnaire consists of 20 items; each item has five numerical response categories (0-4). The total score ranges from 0 to 80, and higher scores are considered to be better functional status. It has been shown to have a sensitive scale to detect changes in functional levels immediately after surgery.
Change from baseline in OBER Test at 6 weeks | [Baseline and 6 weeks]
  The iliotibial tract consists of the fascia lata and the iliotibial band. The iliotibial band is formed by the thickening of the fascia lata lateral to the thigh. The Ober test is used to evaluate Tensor Fascia Lata and iliotibial band tightness. The patient lies in the supine position with the hips and knees extended. The untested leg is brought to abduction, the other leg is moved next to the leg in abduction (hyperadduction). If the Tensor Fascia Lata is short, the leg tested does not go into hyperadduction. In the study conducted by Ferber et al. (2010) regarding the Ober test and iliotibial band flexibility measurements, 300 participants were evaluated with the inclinometer and the average was found to be 24.59 degrees

CONTACTS AND LOCATIONS:
Overall Officials: Ertuğrul Demirdel, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Bayram Sönmez Ünüvar, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No